CLINICAL TRIAL: NCT06528405
Title: The Efficacy and Safety of Sodium-glucose Cotransporter 2 Inhibitors in Patients With Acute Kidney Disease
Acronym: ESS-AKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202404095MINE
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury
Keywords: sodium-glucose cotransporter 2 inhibitor; acute kidney disease; albuminuria
MeSH Terms: conditions — Acute Kidney Injury; Albuminuria | interventions — dapagliflozin; empagliflozin; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGLT2i (Experimental)
  Interventions: Drug: dapagliflozin; Drug: empagliflozin; Drug: canagliflozin
- Control (Placebo Comparator)
  Interventions: Other: Other anti-diabetic drug or no anti-diabetic drug

INTERVENTIONS:
Drug: dapagliflozin — Sodium-glucose cotransporter 2 inhibitor for 90 days during the acute kidney disease period.
  Arms: SGLT2i
Other: Other anti-diabetic drug or no anti-diabetic drug — Other anti-diabetic drug or no anti-diabetic drug for 90 days during the acute kidney disease period.
  Other anti-diabetic drug includes metformin, sulfonylureas, meglitinides, dipeptidyl peptidase-4 inhibitor, insulin, α-glucosidase inhibitors, thiazolidinediones, and glucagon-like peptide-1 receptor agonist.
  Arms: Control
Drug: empagliflozin — Sodium-glucose cotransporter 2 inhibitor for 90 days during the acute kidney disease period.
  Arms: SGLT2i
Drug: canagliflozin — Sodium-glucose cotransporter 2 inhibitor for 90 days during the acute kidney disease period.
  Arms: SGLT2i

SUMMARY:
Acute kidney disease (AKD) happens between 7 and 90 days after an initial kidney injury (AKI). This period is crucial because it can determine whether the condition worsens into chronic kidney disease (CKD). Despite knowing this, there is no proven treatment to improve outcomes for people with AKD.

Recent studies have shown that drugs called sodium-glucose cotransporter 2 (SGLT2) inhibitors can slow down the worsening of chronic kidney disease, help with heart failure, and reduce the risk of death. Now, researchers are looking into whether these drugs can also help prevent acute kidney injury (AKI) and improve outcomes for AKD patients.

Our project will explore the use of SGLT2 inhibitors in patients with AKD, with the belief that these drugs can safely reduce the amount of protein (albumin) in the urine and improve kidney health. To address this, investigators plan to conduct a large, multicenter study in Taiwan. This study will be randomized and placebo-controlled, meaning some patients will receive the SGLT2 inhibitors while others will receive a placebo (a harmless, inactive substance). Investigators will include AKD patients with and without diabetes, focusing on reducing the protein in their urine and monitoring for any serious side effects.

The goal of this trial is to provide strong evidence on whether SGLT2 inhibitors can be an effective treatment for AKD. If successful, this could offer a new strategy to prevent the progression from AKI to CKD and improve the health and outcomes of patients with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 80 years
* Diagnosed with acute kidney disease
* Estimated glomerular filtration rate (eGFR) ≥ 20 mL/min/1.73m²
* Albuminuria > 100 mg/g or proteinuria > 300 mg/g (adjusted by urine creatinine)
* Diagnosed with diabetes or chronic kidney disease

Exclusion Criteria:

* Received sodium-glucose cotransporter 2 (SGLT2) inhibitors within 28 days prior to enrollment
* Patients with type 1 diabetes
* Receiving aggressive immunosuppressive therapy for glomerulonephritis
* Obstructive nephropathy
* Polycystic kidney disease
* Malignancy within 3 months or expected to undergo aggressive treatment such as chemotherapy, radiation therapy, immunotherapy, or targeted therapy in the future
* Pregnant or breastfeeding women
* Clinically assessed as not having recovered from acute kidney injury
* Clinically assessed as at high risk for complications related to SGLT2 inhibitors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Albuminuria | Day 28 and Day 90
  The changes in albuminuria compared with baseline
Discontinuation of SGLT2i | Day 0 to Day 90
  Development of adverse events leading to discontinuation of SGLT2i

SECONDARY OUTCOMES:
eGFR | Day 28 to Day 84 or Day 28 to Day 168
  The changes in eGFR
Major adverse kidney events | Day 0 to Day 180
  eGFR reduction >50%, dialysis, or death
Major adverse cardiovascular events | Day 0 to Day 180
  hospitalization due to heart failure or death
Death | Day 0 to Day 180
  All-cause mortality
Amputation | Day 0 to Day 180
  Any amputation event

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided